CLINICAL TRIAL: NCT05702541
Title: Assessing the Clinical Performance of Two Frequent Replacement Silicone Hydrogel Multifocal Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CLN705-M102
Record Dates: First submitted 2023-01-04; First posted 2023-01-27 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-02

CONDITIONS: Presbyopia
Keywords: Contact lenses
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LID223194 MF, then AOHG MF (Other): Lehfilcon A multifocal contact lenses worn first, followed by lotrafilcon B multifocal contact lenses, as randomized. Each product will be worn in both eyes for 2 days in a daily wear modality. CLEAR CARE will be used for daily cleaning and disinfection.
  Interventions: Device: Lehfilcon A multifocal contact lenses; Device: Lotrafilcon B multifocal contact lenses; Device: Hydrogen peroxide-based cleaning and disinfection system
- AOHG MF, then LID223194 MF (Other): Lotrafilcon B multifocal contact lenses worn first, followed by lehfilcon A multifocal contact lenses, as randomized. Each product will be worn in both eyes for 2 days in a daily wear modality. CLEAR CARE will be used for daily cleaning and disinfection.
  Interventions: Device: Lehfilcon A multifocal contact lenses; Device: Lotrafilcon B multifocal contact lenses; Device: Hydrogen peroxide-based cleaning and disinfection system

INTERVENTIONS:
Device: Lehfilcon A multifocal contact lenses — Silicone hydrogel multifocal contact lenses
  Other Names: LID223194 MF contact lenses
Device: Lotrafilcon B multifocal contact lenses — Silicone hydrogel multifocal contact lenses
  Other Names: AOHG MF contact lenses
Device: Hydrogen peroxide-based cleaning and disinfection system — Commercially available cleaning and disinfection system for silicone hydrogel contact lenses
  Other Names: CLEAR CARE

SUMMARY:
The purpose of this clinical trial is to assess the clinical performance of LID223194 Multifocal (MF) contact lenses and commercially available Air Optix plus HydraGlyde (AOHG) MF contact lenses. Eligible subjects will wear each study lens type in a cross-over fashion as randomized for approximately 2 days.

DETAILED DESCRIPTION:
Subjects will be expected to attend 3 scheduled visits for an individual duration of participation of up to 10 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an consent form (ICF) that has been approved by an Institutional Review Board (IRB);
* Willing to stop wearing habitual contact lenses for the duration of study participation;
* Currently wearing multifocal soft contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months;
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Any eye infection, inflammation, or abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the investigator;
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the investigator;
* History of refractive surgery, or plan to have refractive surgery during the study;
* Current or history of dry eye in either eye that would preclude contact lens wear, in the opinion of the investigator;
* Monovision contact lens wear;
* Other protocol-defined exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (1):
- Johns Creek Research Clinic, Johns Creek, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one investigative site located in the United States.
Pre-assignment Details: This reporting group includes all enrolled participants (16).
Groups:
- LID223194 MF, Then AOHG MF: Lehfilcon A multifocal contact lenses worn first, followed by lotrafilcon B multifocal contact lenses, as randomized. Each product was worn in both eyes for 2 days in a daily wear modality. CLEAR CARE was used for daily cleaning and disinfection.
- AOHG MF, Then LID223194 MF: Lotrafilcon B multifocal contact lenses worn first, followed by lehfilcon A multifocal contact lenses, as randomized. Each product was worn in both eyes for 2 days in a daily wear modality. CLEAR CARE was used for daily cleaning and disinfection.
Period: First Wear Period (Approx 2 Days)
Arm/Group | LID223194 MF, Then AOHG MF | AOHG MF, Then LID223194 MF
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Wear Period (Approx 2 Days)
Arm/Group | LID223194 MF, Then AOHG MF | AOHG MF, Then LID223194 MF
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | LID223194 MF, Then AOHG MF | AOHG MF, Then LID223194 MF | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (3.4) | 60.4 (8.0) | 60.3 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 7 | 12
  Black or African American | 3 | 0 | 3
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Binocular Visual Acuity (VA) With Study Lenses at 4 Meters (logMAR)
Description: VA was assessed binocularly (both eyes together) using a letter chart and measured in logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with lower logMAR values indicating better visual acuity. No hypothesis testing was pre-specified for this endpoint.
Time Frame: Day 2 of each study lens type worn during the corresponding crossover period
Population: This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- LID223194 MF: Lehfilcon A multifocal contact lenses worn during first wear period or second wear period, as randomized.
- AOHG MF: Lotrafilcon B multifocal contact lenses worn during first wear period or second wear period, as randomized.
Arm/Group | LID223194 MF | AOHG MF
Number analyzed (Participants) | 16 | 16
logMAR | -0.06 (0.10) | -0.06 (0.07)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent to study exit, up to 10 days.
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses.
- LID223194 MF Ocular; LID223194 MF Nonocular: Events reported in this group occurred while exposed to the lehfilcon A multifocal contact lenses.
- AOHG MF Ocular; AOHG MF Nonocular: Events reported in this group occurred while exposed to the lotrafilcon B multifocal contact lenses.
Arm/Group | Pretreatment | LID223194 MF Ocular | LID223194 MF Nonocular | AOHG MF Ocular | AOHG MF Nonocular
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/32 | 0/16 | 0/32 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/32 | 0/16 | 0/32 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/32 | 0/16 | 0/32 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT05702541/Prot_SAP_001.pdf